CLINICAL TRIAL: NCT05725954
Title: GUT LINK: A Pilot Study to Evaluate the Comparative Effectiveness of an Evidence-based Care Pathway Across Primary and GI Specialty Care
Brief Title: GUT LINK: A Study of a Care Pathway Across Primary and GI Specialty Care
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Michael Stewart (Other)
Collaborators: Nova Scotia Health Authority (Other)
Responsible Party: Sponsor-Investigator, Michael Stewart, Gastroenterologist, Assistant Professor, Department of Medicine, Dalhousie University, Nova Scotia Health Authority
Organization: Nova Scotia Health Authority (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 50762
Record Dates: First submitted 2023-01-23; First posted 2023-02-13 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Irritable Bowel Syndrome; GI Disorders
Keywords: Care pathway; Care delivery; virtual
MeSH Terms: conditions — Irritable Bowel Syndrome; Digestive System Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GUT LINK SmartPath (Experimental): physicians will use the interactive GUT LINK Smartpath tool in virtual hallway platform to guide their care and referral practices
  Interventions: Behavioral: GUT LINK SmartPath
- control (No Intervention): physicians will provide care and refer as per their usual practices

INTERVENTIONS:
Behavioral: GUT LINK SmartPath — A virtual care delivery and referral support tool for primary healthcare providers.
  Arms: GUT LINK SmartPath

SUMMARY:
It can be challenging for Primary Healthcare Providers (PHCPs) to differentiate between IBS and more serious illnesses involving the GI tract, such as Crohn's disease, ulcerative colitis, or cancer. To help with diagnosis and treatment of IBS, evidence-based guidelines have been developed. However, they are not commonly used in primary care practice and PHCPs and patients often feel that GI specialist evaluation and endoscopy is required. The development of care pathways and clinical practice guidelines is essential to support the investigation and management of digestive diseases, such as IBS.

The current pilot study is designed to assess the implementation and early comparative effectiveness of a Clinical Care Pathway for lower GI tract symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Must be a general practitioner
* Have a family practice in Nova Scotia, Canada
* Utilize the platform 'virtual hallway' as part of current referral practices
* Deliver care to patients with lower GI complaints

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of users | month 3
  Number of users (an indicator of prototype acceptability)
Number of users | month 6
  Number of users (an indicator of prototype acceptability)
Number of referrals | month 3
  Number of referrals from GPs to GI Department (an indicator of prototype acceptability)
Number of referrals | month 6
  Number of referrals from GPs to GI Department (an indicator of prototype acceptability)
Number of referrals per week | month 3
  Number of referrals per week from GPs to GI Department (an indicator of prototype acceptability)
Number of referrals per week | month 6
  Number of referrals per week from GPs to GI Department (an indicator of prototype acceptability)
Number of referrals per user | month 3
  Number of referrals per week from GPs to GI Department (an indicator of prototype acceptability)
Number of referrals per user | month 6
  Number of referrals per week from GPs to GI Department (an indicator of prototype acceptability)
Number of clicks per referral | month 3
  Number of clicks per referral from GPs to GI Department (an indicator of prototype acceptability)
Number of clicks per referral | month 6
  Number of clicks per referral from GPs to GI Department (an indicator of prototype acceptability)
Primary Healthcare Provider Satisfaction | baseline (month 0)
  Thematic analysis of interviews of primary care providers will yield key themes related to satisfaction with the intervention.
Primary Healthcare Provider Satisfaction | month 6
  Thematic analysis of interviews of primary care providers will yield key themes related to satisfaction with the intervention.

SECONDARY OUTCOMES:
Number referrals received as per prototype | month 3
  Number referrals received as per prototype (an implementation metric)
Number referrals received as per prototype | month 6
  Number referrals received as per prototype (an implementation metric)
Number of referrals received requiring troubleshooting | month 3
  Number of referrals received requiring troubleshooting (an implementation metric)
Number of referrals received requiring troubleshooting | month 6
  Number of referrals received requiring troubleshooting (an implementation metric)
Number of referrals aborted | month 3
  Number of referrals aborted (an implementation metric)
Number of referrals aborted | month 6
  Number of referrals aborted (an implementation metric)
Type of consult | month 3
  Type of consult (Full consult, specialist telephone advice, eConsult)
Type of consult | month 6
  Type of consult (Full consult, specialist telephone advice, eConsult)
Perceived appropriateness of the SmartPath | month 3
  Thematic analysis of interviews of primary care providers will yield key themes related to the perceived appropriateness of the intervention
Perceived appropriateness of the SmartPath | month 6
  Thematic analysis of interviews of primary care providers will yield key themes related to the perceived appropriateness of the intervention
physician self-efficacy rating | month 3
  physician self-efficacy rating, measured using the 'New General Self Efficacy Scale' (an effectiveness metric of GUT LINK Smartpath). Min score: 1, max score: 8. A higher score indicates a greater self-efficacy.
physician self-efficacy rating | month 6
  physician self-efficacy rating, measured using the 'New General Self Efficacy Scale' (an effectiveness metric of GUT LINK Smartpath). Min score: 1, max score: 8. A higher score indicates a greater self-efficacy.
Referral triage priority category | month 3
  Referral triage priority category will be collected from referrals through the pathway (an effectiveness metric of GUT LINK Smartpath). Referral triage categories to the GI department are: emergent, semi urgent, and non-urgent.
Referral triage priority category | month 6
  Referral triage priority category will be collected from referrals through the pathway (an effectiveness metric of GUT LINK Smartpath). Referral triage categories to the GI department are: emergent, semi urgent, and non-urgent.
Time from referral to specialist consultation | month 3
  Time from referral to specialist consultation, in weeks (an effectiveness metric of GUT LINK Smartpath)
Time from referral to specialist consultation | month 6
  Time from referral to specialist consultation, in weeks (an effectiveness metric of GUT LINK Smartpath)
Time from referral to diagnosis and treatment | month 3
  Time from referral to diagnosis and treatment, in weeks (an effectiveness metric of GUT LINK Smartpath)
Time from referral to diagnosis and treatment | month 6
  Time from referral to diagnosis and treatment, in weeks (an effectiveness metric of GUT LINK Smartpath)

CONTACTS AND LOCATIONS:
Locations (1):
- QEII Health Sciences Centre, Halifax, Nova Scotia, Canada